CLINICAL TRIAL: NCT03806335
Title: The Effect of Local Infiltration Technique on Postoperative Pain After Adult Tonsillectomy: A Randomized Double-blind Clinical Trial
Brief Title: The Effectiveness of Local Infiltration Technique in Adult Tonsillectomy
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of patients
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Zoher Naja, Anesthesiologist, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 32015
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infiltration (Experimental): Patients will receive pre-incision infiltration of 2.5 ml local anesthesia mixture in each tonsil.
  Interventions: Other: Infiltration; Other: General anesthesia
- Placebo (Placebo Comparator): Patients will receive pre-incision infiltration of 2.5 ml saline in each tonsil.
  Interventions: Other: Placebo; Other: General anesthesia

INTERVENTIONS:
Other: Infiltration — The infiltration will be performed by the anesthetist using a 25G- 3.5cm curved needle. A total of 2.5 ml of local anesthetic mixture will be used for each tonsil. The mixture will contain: 10 ml xylocaine 2% an d10 ml bupivacaine 0.5%
  Arms: Infiltration
Other: Placebo — Patients will receive 2.5 ml normal saline in each tonsil
  Arms: Placebo
Other: General anesthesia — All patients will receive general anesthesia prior to infiltration

SUMMARY:
Tonsillectomy is commonly associated with postoperative pain. The modified pre-incision infiltration of anesthetic mixture combined with general anesthesia was shown to decrease post-tonsillectomy pain in children. Hence, the present clinical trial will assess the effectiveness of this technique in adults undergoing tonsillectomy.

DETAILED DESCRIPTION:
The study will be conducted prospectively, using a randomized double-blind design. Adult patients scheduled for total or partial tonsillectomy with or without adenoidectomy starting from January 2019 till January 2020 will be included.Patients will be allocated randomly into two equal groups using the sealed envelope method. Both groups will receive general anesthesia. Then, one group will receive pre-incision infiltration of 2.5 ml local anesthesia mixture in each tonsil. The second group will have placebo infiltration.

ELIGIBILITY:
Inclusion Criteria:

* patients with total or partial tonsillectomy with or without adenoidectomy

Exclusion Criteria:

* patients who took antiemetics, steroids, or antihistaminics within 24 hours before surgery. - patients who have asthma
* patients who have diabetes
* patients who have bleeding problems
* patients who are suspected to have signs of acute pharyngeal infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Post operative pain | within 10 days after the operation
  Pain after the operation will be assessed using the Visual Analogue Scale (VAS). A minimum VAS score is 0 and the maximum score is 10.

SECONDARY OUTCOMES:
PONV | within 10 days after the operation
  Post operative nausea and vomiting (PONV) will be assessed through a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Zoher Naja, Principal Investigator — Makassed General Hospital
Locations (1):
- Makassed General Hospital, Beirut, Lebanon